CLINICAL TRIAL: NCT02390947
Title: A Multicenter，Randomized, Double-blind, Placebo-controlled Trial of Famitinib in Patients With Advanced Colorectal Adenocarcinoma
Brief Title: Safety and Efficacy Study of Famitinib in Patients With Advanced Colorectal Adenocarcinoma（FACT）
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-FMTN-CRC-FACT
Record Dates: First submitted 2015-02-26; First posted 2015-03-18 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Recurrent
Keywords: Colorectal Cancer; Famitinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — famitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Famitinib arms (Experimental): Famitinib 25 mg p.o. qd and the medication continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Famitinib
- Control arms (Placebo Comparator): Placebo 25 mg p.o. qd and the medication continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famitinib — 25 mg p.o. qd
  Arms: Famitinib arms
Drug: Placebo — 25 mg p.o. qd
  Arms: Control arms

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3, whose anti-tumor and anti-angiogenesis effects have been validated in preclinical tests. In PhaseⅡb study, a significantly improved Progression Free Survival (PFS) was found in patients with advanced colorectal cancer treated with Famitinib compared to placebo. On the other hand, the toxicity of Famitinib was manageable in both PhaseⅠand Ⅱb studies.

The purpose of this study is to determine whether Famitinib can improve Overall Survival (OS) compared with placebo in total 540 patients with advanced colorectal cancer who have failed in previously received at least two lines of standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 75 (including 18 and 75) at the time of Informed Consent
2. Pathologically confirmed advanced colorectal adenocarcinoma (all the other histological types are excluded)
3. Treatment failure in previously received standard therapy (at least two lines), which must include 5-Fu, irinotecan and oxaliplatin

   Definition of "treatment failure":

   A.Disease progression during experimental drug treatment or within 3 months after the last treatment, with definite imaging or clinical evidences;

   B.For patients abandoning chemotherapy because of intolerance of advent events, hematologic toxicity is required to reach ≥Grade IV (platelet decrease ≥ Grade III ), and nonhematologic toxicity is required to reach ≥Grade III , according to NCI CTCAE 4.0. Furthermore, the original treatment should be not tolerated any more when it is repeated to the same patient, judged by investigators.

   Note:

   A.When adjuvant therapy including oxaliplatin was previously used, at least 9 courses of FOLFOX (2 weeks regimens), 6 courses of CapeOX (3 week regimen), or 750mg/m^2 cumulative consumption of oxaliplatin, are required. Adjuvant therapy will be regarded as the first-line treatment when disease progressed during or within 6 months after treatments

   B.Monoclonal antibody drugs (bevacizumab, cetuximab, panitumumab, aflibercept, etc.) are allowed to combine with prior chemotherapy.
4. At least one measurable targeting lesion according to RECIST 1.1 (The diameter of tumor and lymph node lesion should be ≥ 10 mm and 15mm, respectively, with scanning layer ≤ 5 mm and without local treatment)
5. Eastern Cooperative Oncology Group (ECOG) performance status:0-1.
6. Life expectancy ≥ 3 months
7. Adequate function of major organs, meaning the following criteria should be met within 14 days before randomization:

   A.Routine blood test:
   1. Hemoglobin > 90g/L (not received blood transfusion or drugs to incraese RBC, Hb, WBC and PLT in 14 days before screening )
   2. Neutrophils > 1.5×10^9/L
   3. Platelets > 100×10^9/L

      B. Blood biochemistry:
   4. Total bilirubin < 1.25×the upper limit of normal (ULN)
   5. Serum transaminase ≤ 2×ULN (≤ 5×ULN, If existing liver metastases)
   6. Creatinine clearance rate ≥ 60ml/min (Cockcroft-Gault Formula)

   C.Doppler echocardiography assessment: Left ventricular ejection fraction (LVEF) ≥ 50%
8. Having recovered from impairments of other therapy before taking research drugs (more than 6 weeks from the last treatment of Nitroso or MMC, more than 4 weeks from the last treatment of other cytotoxic drugs, targeted drugs, radiotherapy or operation, with completely healed wound, more than 2 weeks from the last treatment of Chinese traditional and patent medicine)
9. Signed and dated informed consent
10. Good compliance of patients and agreement of their family members to cooperate on the follow-up of survival.

Exclusion Criteria:

1. Second malignancies, except for cured skin basal cell carcinoma and carcinoma in-situ of uterine cervix, before or during screening
2. Previously received therapy of tyrosine kinase inhibitor agent targeting at VEGFR, e.g. famitinib, sorafenib, sunitinib, regorafenib
3. Having joined in other clinical trials within 4 weeks
4. Factors influencing the usage of oral administration (e.g. unable to swallow, chronic diarrhea and intestinal obstruction, etc.)
5. Having haemorrhage history, ≥ Grade Ⅲ (NCI CTCAE 4.0 ) haemorrhage occurred within 4 weeks before screening
6. Known central nervous system (CNS) metastasis or having CNS metastasis history before screening. CT or MRI scan should be received 28 days before randomization when CNS metastases is clinically suspected
7. Uncontrolled hypertension with single medical therapy (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), History of unstable angina pectoris or newly diagnosed unstable angina pectoris within 3 months before screening, myocardial infarction events within 6 months before screening, Arrhythmias (QTcF: ≥450ms in male, ≥ 470ms in female) needed long-term treatment of drugs, ≥ class II cardiac insufficiency by New York Heart Association (NYHA) classification
8. urinary protein ≥ ++ or 24-hour urinary protein ≥ 1.0 g
9. Chronic untreated wounds or fractures
10. Tumor invasion around major vessels shown by imaging, high risk of major vascular invasion leading to massive hemorrhage judged by investigators
11. Abnormal international normalized ratio (INR) of patients with coagulation dysfunction and hemorrhagic tendency at 14 days before randomization. Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues. However, low doses of warfarin (1mg orally, once daily) or aspirin (between 80mg to 100mg daily) can be used for prevention on the premise of INR ≤ 1.5
12. Artery/venous thromboembolic events occurred within 1 year before screening, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis (except for recovered venous thrombosis judged by investigators, which was caused by venous catheter in previous chemotherapy) and pulmonary embolism, etc.
13. All female patients who are not surgically sterilized or postmenopausal refusing to take a reliable method of birth control during the study and within 6 months after the last dose of test article. All female patients in breastfeeding period or in child-bearing period with a positive urine or serum pregnancy test result before randomization. All male subjects who are not surgically sterilized refusing to take a reliable method of birth control during the study and within 6 months after the last dose of test article.
14. Preexisted thyroid dysfunction, thyroid function cannot be controlled within normal range even using medical therapy
15. History of psychiatric drug abuse and addiction, dysphrenia
16. Symptomatic pleural effusion, hydropericardium or ascites needed clinical intervention or being stable less than 4 weeks.
17. History of Immunodeficiency, acquired or congenital immunodeficiency, history of organ transplantation
18. Known active HBV or HCV infection companion with hepatic dysfunction
19. Concomitant disease judged by investigators that may bring serious harm to the safety of patients or the completion of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival(OS) | 3 years

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 1.5 years
Objective response rate(ORR) | 6 months
Disease Control Rate(DCR) | 1.5 years
Quality of Life as measured by EORTC QLQ-C30(3.0) | 1.5 years
The incidence of Adverse Events | 3 years
The severity of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, M.D, Principal Investigator — Beijing Cancer Hospital, Peking University; Ruihua Xu, M.D, Principal Investigator — Cancer Center, Sun Yet-sen University
Locations (44):
- China (44):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Peking University, Beijing, Beijing Municipality
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - PLA Hospital 301, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of The Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Cancer center, Sun Yet-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University of Chinese Medicine, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Hainan, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The first affiliated hospital of Xinxiang medical university, Xinxiang, Henan
  - Cancer Hospital of Henan Province, Zhengzhou, Henan
  - The First affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - Cancer Hospital of Hunan Province, Changsha, Hunan
  - The Third Xiangya Hospital of Cental South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Cancer Hospital of Jiangsu Province, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical Collage, Xuzhou, Jiangsu
  - Cancer Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Cancer Hospital of Jilin province, Changchun, Jilin
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Cancer Hospital of Liaoning Province, Shenyang, Liaoning
  - Chinese Medical University First Hospital, Shenyang, Liaoning
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai jiaotong University, School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Cancer Hospital of Shanxi Province, Xian, Shanxi
  - Tangdu Hospital of The Fouth Military Medical University, Xian, Shanxi
  - Cancer Hospital of Tianjin City, Tianjin, Tianjin Municipality
  - People's Hospital of Tianjin City, Tianjin, Tianjin Municipality
  - Cancer Hospital of Yunnan Province, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang